CLINICAL TRIAL: NCT05231746
Title: A Phase 1, Multicenter, Open-label Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of hSTC810 Monotherapy in Subjects With Advanced Solid Tumors
Brief Title: A Study of hSTC810 With Advanced/Metastatic Solid Tumors (STCUBE-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: STCube, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STCUBE-001
Record Dates: First submitted 2022-01-25; First posted 2022-02-09 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor
Keywords: Immune Checkpoint Inhibitors; Antineoplastic Agents; Therapeutic Uses; Colorectal Neoplasms; Head and Neck Neoplasms; Ovarian Neoplasms; Urinary Bladder Neoplasms; Lung Neoplasms; Antibodies, Monoclonal; anti-BTN1A1; butyrophilins
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Ovarian Neoplasms; Urinary Bladder Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- hSTC810 (Experimental): 6 escalating doses of hSTC810 will be administered to participants
  Interventions: Biological: hSTC810

INTERVENTIONS:
Biological: hSTC810 — hSTC810 will be administered as an intravenous infusion (IV)

SUMMARY:
The Purpose of this study is to investigate the safety, tolerability, pharmacokinetics, and preliminary efficacy of hSTC810 monotherapy in participants with advanced solid tumors.

DETAILED DESCRIPTION:
The study consists of a dose-escalation phase that will evaluate 6 dosing schedules of hSTC810. The first cohort will be single participant cohort. Subsequent escalation cohorts will use a standard 3+3 design, with the ability to backfill up to an additional 6 patients in each dose cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged at 18 ≥ years
* Capable and willing to give signed informed consent
* At least one measurable lesion as determined by RECIST Ver.1.1
* ECOG PS score ≤ 1
* Expected survival ≥ 12 weeks
* For female or male patients of reproductive potential: Agree to use contraception throughout the study and at least 6 months after the last dose.

Exclusion Criteria:

* Subject who has received anti-cancer treatment within 4 weeks prior to the first dose of study treatment.
* Subject who has received radiotherapy or major surgery within 4 weeks prior to screening.
* Any toxicity due to prior therapy that has not resolved to ≤ Grade 1 or returned to baseline by the time of starting study treatment.
* Subject with known severe (≥Grade 3) hypersensitivity to any checkpoint inhibitor.
* Clinically significant laboratory abnormalities.
* Subject with a history of another invasive malignancy within 3 years before the first dose of study drug.
* Subject with active central nervous system (CNS) metastases.
* Subject who requires high dose of steroids or other immunosuppressive medications.
* Subject with a history of autoimmune disease that has required systemic treatment in the past 2 years.
* Subject with active infection that requires systemic antimicrobial treatment.
* Subject with active HBV or HCV infection.
* Subject who has a known history of HIV infection.
* Subject with active tuberculosis.
* Subject with a documented history of a cerebral vascular event, unstable angina, myocardial infarction, or cardiac symptoms consistent with NYHA Class IV within 6 months prior to screening.
* Subject with a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening CT scan.
* Subject who has received a prior allogeneic stem cell or solid organ transplant.
* Subject with a positive coronavirus disease (COVID) test during screening.
* Subjects who have received a live attenuated vaccine within 30 days prior to screening.
* Subject with another underlying medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs | 4 weeks
  Number and percentages of subjects with DLTs
Incidence of AEs, SAEs, and abnormalities in Lab | from signing ICF to 90 days after last dose
  Number and percentages of subjects with Adverse Event, serious AEs, and abnormalities in lab parameters

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Up to 2 years
  Maximum plasma concentration of hSTC810 to evaluate the PK parameters
Minimum plasma concentration (Cmin) | Up to 2 years
  Minimum blood plasma concentration of hSTC810 to evaluate the PK parameters
Time to maximum plasma concentration (Tmax) | Up to 2 years
  Time to reach Cmax of hSTC810 to evaluate the PK parameters.
Area under the plasma concentration - time curve (AUC0-t) | Up to 2 years
  AUC up to the last measurable concentration of hSTC810 to evaluate the PK parameters
Incidence of ADA | Up to 2 years
  Number and percentages of subjects with positive ADAs
Objective response rate (ORR) | Up to 2 years
  Percentage of participants with confirmed CR and confirmed PR determined by RECIST v1.1 and iRECIST
Best overall response (BOR) | Up to 2 years
  the best response designation as determined by RECIST and iRECIST. The BOR will be categorized as a CR, PR, SD, or PD
Clinical Benefit rate (CBR) | Up to 2 years
  Percentage of Participants With confirmed CR, confirmed PR or SD with a duration of at least 6 months determined by RECIST v1.1 and iRECIST
Duration of response (DoR) | Up to 2 years
  Time from initial response of confirmed CR or PR to disease progression or death determined by RECIST v1.1 and iRECIST
Progression free survival (PFS) | Up to 2 years
  The period from the first dose to the documented disease progression or death determined by RECIST v1.1 or iRECIST
Overall survival (OS) | Up to 2 years
  The period from first dose to the day of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical director, Study Director — STCube, Inc.
Locations (5):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - Mount Sinai Hospital, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- South Korea (2):
  - Korea University Anam Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No